CLINICAL TRIAL: NCT02953171
Title: A Randomized Controlled Clinical Trial to Investigate the Efficacy of Lacto-fermented Sauerkraut and the Probiotic E. Coli Nissle 1917 in the Treatment of Irritable Bowel Syndrome
Brief Title: Probiotics in the Treatment of Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Eirik Garnås, Public Health Nutritionist, University of Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/1129/REK
Record Dates: First submitted 2016-10-17; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; The human microbiome; Microbiota; Gut microbiota; Probiotics; Sauerkraut
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Airway Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Raw sauerkraut+Probiotic capsule (Experimental): 75 grams of raw, lacto-fermented sauerkraut + 1 capsule of the probiotic Mutaflor, each day for 6 weeks.
  Interventions: Other: Raw, lacto-fermented sauerkraut; Dietary Supplement: Mutaflor
- Raw sauerkraut+placebo capsule (Experimental): 75 grams of raw, lacto-fermented sauerkraut + 1 placebo capsule, each day for 6 weeks.
  Interventions: Other: Raw, lacto-fermented sauerkraut; Other: Placebo capsule
- Pasteurized sauerkraut+Probiotic capsule (Experimental): 75 grams of pasteurized sauerkraut + 1 capsule of the probiotic Mutaflor, each day for 6 weeks.
  Interventions: Dietary Supplement: Mutaflor; Other: Pasteurized sauerkraut
- Pasteurized sauerkraut+Placebo capsule (Placebo Comparator): 75 grams of pasteurized sauerkraut + 1 placebo capsule, each day for 6 weeks.
  Interventions: Other: Pasteurized sauerkraut; Other: Placebo capsule

INTERVENTIONS:
Other: Raw, lacto-fermented sauerkraut — Sauerkraut fermentations have been shown to contain a broad range of microorganisms, including Leuconostoc mesenteroides, Lactobacillus plantarum, Leuconostoc citreum, Leuconostoc argentinum, Lactobacillus paraplantarum, and Lactobacillus coryniformis. Some of these bacteria, such as Lactobacillus plantarum, are classified as probiotics.
  Arms: Raw sauerkraut+Probiotic capsule; Raw sauerkraut+placebo capsule
Dietary Supplement: Mutaflor — The probiotic Escherichia coli Nissle 1917, registered in Germany as the medicinal product Mutaflor, possesses a unique combination of fitness and survival factors.
  Arms: Pasteurized sauerkraut+Probiotic capsule; Raw sauerkraut+Probiotic capsule
Other: Pasteurized sauerkraut — Sauerkraut without live bacteria.
  Arms: Pasteurized sauerkraut+Placebo capsule; Pasteurized sauerkraut+Probiotic capsule
Other: Placebo capsule — Capsules without probiotics
  Arms: Pasteurized sauerkraut+Placebo capsule; Raw sauerkraut+placebo capsule

SUMMARY:
The aim of the present study is to assess the efficacy of two different probiotic products, lacto-fermented sauerkraut and the supplement Mutaflor, in the treatment of irritable bowel syndrome.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic gastrointestinal (GI) disorder that affects around 11% of the population globally. Several factors have been implicated in the pathogenesis of IBS, including psychological stress, gastrointestinal motility, and diet. More recently, it has become clear that the gastrointestinal microbiota may play a critical role in the pathophysiology of this functional GI condition.

Gut microbiome manipulation, for example through the use of probiotic and prebiotic supplements, has shown some promise in the treatment of IBS. However, the research in this area is still in its infancy, and it remains unclear what type of intervention that is the preferred choice in cases of IBS. Many, if not most, probiotic supplements on the market today contain bacteria that are incapable of colonizing the human gut, which may partly explain why the health effects associated with the use of probiotics tend to be temporary, rather than permanent.

Several studies have investigated how the use of probiotic supplements containing Bifidobacteria and Lactobacilli affect the clinical outcome of patients with IBS. However, to date, no studies have assessed whether fermented vegetables, a "natural" source of probiotic bacteria, are useful in the treatment of IBS. Moreover, little is known about how other types of probiotic bacteria, such as those belonging to the genus Escherichia, affect symptoms of IBS.

ELIGIBILITY:
Inclusion Criteria:

Rome III criteria (Criteria fulfilled for the last 6 months with symptom onset at least 3 months prior to diagnosis):

Recurrent abdominal pain or discomfort at least 3 days/month in the last 3 months associated with two or more of the following:

1. Improvement with defecation
2. Onset associated with a change in frequency of stool
3. Onset associated with a change in form (appearance) of stool

Exclusion Criteria:

* Psychiatric disorder
* Metabolic disease
* Chronic infection
* Organic gastrointestinal disorder
* Pregnancy
* Breastfeeding

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
IBS Symptom Severity Scale (IBS-SSS). | Change from day 0 to day 42

SECONDARY OUTCOMES:
Body weight | Change from day 0 to day 42
Fecal microbiome diversity | Change from day 0 to day 42
  16S rRNA gene sequences (prokaryotes)
The Quality of Life Scale (QOLS) | Change from day 0 to day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Volvat Medisinske Senter, Majorstuen, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided